CLINICAL TRIAL: NCT02505321
Title: Defining Adipose Tissue Lipid Deposition in Normal Weight Individuals With a Genetic Predisposition to Insulin Resistance
Brief Title: for Adipose Tissue DIabetes VAriants (fATDIVA)
Acronym: fATDIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CRF 180; 1508127 (Other: Royal Devon & Exeter NHS Foundation Trust R&D)
Record Dates: First submitted 2015-07-06; First posted 2015-07-22 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus
Keywords: insulin resistance; physiology; genetics; gene variants; pathogenesis; type 2 diabetes; fat; polygenic lipodystrophy
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 2; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fATDIVA - OTTT (Cases) (Experimental): Individuals identified with the "polygenic lipodystrophy" genetic variants of interest will undergo the Oral Triglyceride Tolerance Test (OTTT) plus an abdominal fat biopsy (optional). Case/control status will be unblinded at analysis.
  Interventions: Other: Oral Triglyceride Tolerance Test (OTTT); Procedure: Abdominal fat biopsy (optional)
- fATDIVA - OTTT (Controls) (Experimental): Control individuals carrying the average number of risk alleles and matched to individuals identified with the "polygenic lipodystrophy" genetic variants of interest for gender, age and BMI, will undergo the Oral Triglyceride Tolerance Test (OTTT) plus an abdominal fat biopsy (optional). Case/control status will be unblinded at analysis.
  Interventions: Other: Oral Triglyceride Tolerance Test (OTTT); Procedure: Abdominal fat biopsy (optional)

INTERVENTIONS:
Other: Oral Triglyceride Tolerance Test (OTTT) — Participants consume a fatty drink. An intravenous catheter is inserted into the antecubital veins in one arm for intermittent sampling over the following 4 hours. The OTTT permits simple evaluation of postchallenge triglyceride levels and is acceptable to participants.
  Other Names: OTTT
Procedure: Abdominal fat biopsy (optional) — A sample of abdominal fat will be obtained by firstly injecting some local anaesthetic into an accessible area of the abdomen. Using a scalpel, a small incision (approx 2-3 cm) will be made to a depth of approx 15mm and two small pea-sized samples of fat will be removed. The wound will be closed with simple sutures or steristrips.

SUMMARY:
The adipose (fat) cells under the skin are where individuals store excess fat. The more excess fat they have, the more "strain" they put on these cells which then get bigger and don't work as well as they should. Having some fat under the skin is important. People who have a genetic defect which results in them having almost no fat under their skin have a very high risk of a condition called insulin resistance (where the body does not respond as well to insulin and blood sugar levels rise). This can lead to diabetes and heart disease despite them not being overweight.

Scientists have only recently started to understand the importance of fat in insulin resistance and how people unable to store fat very well can have insulin resistance despite not being obese. The investigators have also recently discovered that small changes in a person's genetic code (their body's instruction manual) may also affect their ability to store fat and would like to explore this in more detail. To do this, they will recruit volunteers from the Exeter 10,000 study who gave permission to contact them about further research. The investigators will collect detailed body size measures and blood samples taken before and after a special drink that is high in fat (similar to a thick milk shake), then compare the results between people with and without the particular genetic changes of interest.

Knowing more about these genetic changes and how fat cells work could help to improve understanding about why some people develop diabetes and heart disease despite a relatively normal BMI.

DETAILED DESCRIPTION:
Hypothesis:

Individuals carrying different genetic variations have different abilities to store fat under the skin.

Aim: To improve understanding of "adipose tissue dysfunction" using human genetics, and demonstrate that lipid uptake into fat cells is compromised in subjects with 'polygenetic lipodystrophy' alleles.

Objectives:

* Identify individuals with genetic risk variants of interest and controls matched for gender, age and BMI.
* Undertake detailed physiological assessments including an Oral Triglyceride Tolerance Test (OTTT) (blood samples before and after a fatty drink), detailed body size measures and an optional fat biopsy.
* Using the samples collected, test whether or not individuals carrying a high genetic load of "polygenic lipodystrophy" alleles:

  1. have larger subcutaneous fat cells.
  2. have higher circulating lipid levels 4 hours after a fatty meal challenge.
  3. have a gene expression profile normally associated with obesity, despite being of the same BMI as matched controls. This profile includes a downregulation of genes involved in fatty acid trafficking and an upregulation of genes involved in inflammation.
  4. have higher insulin resistance as measured by HOMAIR (calculated from fasting insulin and fasting glucose).

Background:

Diabetes is the most common chronic metabolic disease and is a major source of morbidity and mortality. It is one of the biggest healthcare challenges facing the UK NHS with more than 2.6 million adults diagnosed in the UK, with the vast majority (90%) having type 2 Diabetes (T2D). It is anticipated the numbers will continue to rise, in part due to the increasing levels of obesity in the population.

T2D is characterised by high blood glucose levels in the context of increasing insulin resistance and reduced beta cell function, and this can develop over several years with individuals unaware of the problem.

Research groups in Exeter are leading efforts to identify the genetic factors that influence why some people develop T2D despite relative leanness, whilst many obese people do not get the disease. The investigators have identified many such factors but now wish to study them in more detail to understand the role of insulin.

Introduction:

Adipose tissue dysfunction Working with collaborators as part of ongoing genetic studies, the investigators have identified several genetic variations (DNA changes) associated with insulin resistance, and believe some of these genetic variants operate primarily through adipose tissue "dysfunction". Adipose tissue dysfunction is a relatively new concept and has resulted from detailed physiological studies that have revealed that obese individuals have larger fat cells, more inflamed fat tissue (often infiltrated with macrophages) poorer adipose tissue blood flow pre/post meal, and differential expression of genes involved in these processes (Alkhouli 2013). The failure of adipocytes, resulting in a limited capacity to take up free fatty acids (FFA), predispose to ectopic fat depositions which is a deposition of lipids in sites such as the liver, muscle with more omental tissue similar to subjects with lipodystrophy.

The investigators are trying to understand how genetic variations cause differences in people's ability to store fat and wish to test the hypothesis that individuals carrying different genetic variations have different abilities to store fat under the skin as subcutaneous fat tissue. This could lead to an improved understanding of subcutaneous fat storage. It is very unlikely that the rising numbers of people becoming overweight or obese as they age will be substantially reversed, therefore the study's findings could be important in identifying how to reduce the risk of disease caused by obesity.

Methods:

Study design:

This is a prospective "recruit by genotype" cohort study that will take place over a 2 year period (2015 to 2017).

Study participants:

All participants will be identified from existing research cohorts managed by the NIHR Exeter Clinical Research Facility (Exeter CRF) and recruitment will be facilitated within the Exeter CRF.

Under over-arching ethical approval 09/H0106/75, approximately 7500 anonymised DNA samples have been genotyped for genetic variants related to insulin production. These variants occur in >1% of the population and have no direct consequences to individual health.

There is no defined cut-off for having, or not having, polygenic lipodystrophy as it is not based on a single genetic variant. People will have between 0 and 22 polygenic lipodystrophy alleles and the investigators are looking for those with a combination of at least 11 genetic variants. They have identified approx 300 people in the EXTEND cohort who fit this criteria and will then recruit matched controls from those in the EXTEND cohort who have been identified as having the fewest number of risk alleles.

Recruitment:

The investigators will provide the Exeter Clinical Research Facility (Exeter CRF) with a list of the sample numbers that have been identified as having the Individuals identified with the "polygenic lipodystrophy" genetic variants of interest, together with control individuals carrying the average number of risk alleles. The Exeter CRF Data Manager will then identify 50 individuals with the variants and 50 individuals matched for age, gender, diabetes status and BMI, who will be invited to a 5-hour visit to the Exeter CRF for data and sample collection. Interested participants will be contacted directly by a member of the study team who will be responsible for the recruitment process, providing more detailed verbal and written project-specific information.

Procedure:

All participants will be asked to refrain from strenuous exercise and from eating very fatty meals in the 48 hours prior to coming in to the clinic, and no alcohol (it has high energy content and affects the liver) but otherwise normal diet, then fast overnight prior to attending a morning visit at the Exeter CRF. Participants will be asked to sign a written consent form prior to any data collection.

Data collection:

Anthropometry:

* Baseline data including Ht (m), Wt (kg), Waist (cm) and Hip (cm) circumference will be recorded.
* Detailed body fat measures will be obtained from the BOD POD.
* Skin fold measurements (mm) from biceps, triceps, subscapular, and suprailiac regions.

Medical history: including current medications and lifestyle information (smoking/alcohol).

BODPOD TM :

Detailed body composition measures will be obtained using the Body Composition Tracking System. This briefly comprises a BOD POD machine, electronic scales, and a computer. It uses the principles of body densitometry (measuring mass and volume) to calculate the participant's percentage and absolute amounts of fat and fat free mass. Participants will be asked to wear minimal clothing (e.g. swimming costume) and a close fitting swim hat. They stand on the electric scales to record their weight which is then calibrated with the BOD POD. Participants are asked to sit inside the BOD POD up to 1 minute at a time (max 3 times). The computer will then analyse and generate the results.

Blood samples:

Oral Triglyceride Tolerance Test (OTTT) (approx. 4 hours):

A small cannula (thin plastic tube) will be inserted into a vein following standard clinical practice to minimize any potential trauma from repeat blood sampling.

* Fasting samples (at -5 and -2 minutes) will be obtained for baseline measures (including routine glucose and lipid measurement) plasma and serum for storage and future batched analysis, and pre-OTTT measures of glucose, insulin, standard lipids, and stored plasma for potential future metabolomic or lipidomic studies.
* Following the initial fasting blood sampling, the participant will be asked to drink approx 150 mls of Fresubin 5cal shot supplement drink over a 5 min period. The time of completion will be noted as T= 0. Further blood samples will be obtained at T=30, 60, 120, 180 and 240 minutes post-ingestion. The calorific content and proportion of macronutrients in Fresubin is very similar to that described in publications performing the OTTT (Karamanos 2001; Carstensen 2003; Mohanlal 2004).

At the end of this period the cannula will be removed and the participant will be offered a light lunch/refreshments.

Optional abdominal fat biopsies (approx. 30 mins and undertaken during OTTT):

For research volunteers that are happy to undergo a small fat biopsy, a sample of abdominal fat will be obtained by firstly injecting some local anaesthetic into an accessible area of the abdomen. Using a scalpel, a small incision (approx 2-3 cm) will be made to a depth of approx 15mm and two small pea-sized samples of fat will be removed. The wound will be closed with simple sutures or steristrips. One fat sample will be flash frozen in liquid nitrogen immediately after excision and stored at minus 80 degrees for RNA analyses. The other sample will be stored in formalin for later immunohistochemistry staining.

ELIGIBILITY:
Inclusion Criteria:

* Demographics: Age 18-75 inclusive
* Ethnicity: Reflective of local demographic
* Mental capacity: Willing and able to provide informed consent

Exclusion Criteria:

* Medical history: Treated Diabetes (including insulin and GLP-1 analogues), history of bariatric surgery and recent significant weight loss/gain (+/- 3 kgs/half a stone in the last 3 months); connective tissue disease, pregnancy and lactation.
* Medications: Currently prescribed glucose-lowering medication (we will NOT exclude those controlling their diabetes with diet alone), oral/IV corticosteroid treatment or loop diuretics (furosemide, bumetanide), antiplatelet and anticoagulation medication, methotrexate
* Mental capacity: Unable/unwilling to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Level of Circulatory Lipids following Triglyceride stimulation test (OTTT) (mmol/L) | Within 12 months of recruitment date of final participant
  Level of Circulatory Lipids will be assessed using measures of triglyceride levels from each post-prandial time point sample.

SECONDARY OUTCOMES:
Mean adipocyte size assessed using Image J | Within 12 months of recruitment date of final participant
  ImageJ is a cross-platform image analysis tool developed to measure particle/cell size and will be used here to measure adipocyte size.
Incremental Area under the Curve NEFA levels (µmol/L) | Within 12 months of recruitment date of final participant
  Incremental Area under the Curve NEFA levels, calculated using values/levels from each post-prandial sample time point and subtracting fasting values.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Frayling (Prof), PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaghootkar H, Scott RA, White CC, Zhang W, Speliotes E, Munroe PB, Ehret GB, Bis JC, Fox CS, Walker M, Borecki IB, Knowles JW, Yerges-Armstrong L, Ohlsson C, Perry JR, Chambers JC, Kooner JS, Franceschini N, Langenberg C, Hivert MF, Dastani Z, Richards JB, Semple RK, Frayling TM. Genetic evidence for a normal-weight "metabolically obese" phenotype linking insulin resistance, hypertension, coronary artery disease, and type 2 diabetes. Diabetes. 2014 Dec;63(12):4369-77. doi: 10.2337/db14-0318. Epub 2014 Jul 21. PMID 25048195
- [Background] Semple RK, Sleigh A, Murgatroyd PR, Adams CA, Bluck L, Jackson S, Vottero A, Kanabar D, Charlton-Menys V, Durrington P, Soos MA, Carpenter TA, Lomas DJ, Cochran EK, Gorden P, O'Rahilly S, Savage DB. Postreceptor insulin resistance contributes to human dyslipidemia and hepatic steatosis. J Clin Invest. 2009 Feb;119(2):315-22. doi: 10.1172/JCI37432. Epub 2009 Jan 26. PMID 19164855
- [Background] Stears A, O'Rahilly S, Semple RK, Savage DB. Metabolic insights from extreme human insulin resistance phenotypes. Best Pract Res Clin Endocrinol Metab. 2012 Apr;26(2):145-57. doi: 10.1016/j.beem.2011.09.003. PMID 22498245
- [Background] Alkhouli N, Mansfield J, Green E, Bell J, Knight B, Liversedge N, Tham JC, Welbourn R, Shore AC, Kos K, Winlove CP. The mechanical properties of human adipose tissues and their relationships to the structure and composition of the extracellular matrix. Am J Physiol Endocrinol Metab. 2013 Dec;305(12):E1427-35. doi: 10.1152/ajpendo.00111.2013. Epub 2013 Oct 8. PMID 24105412
- [Background] Karamanos BG, Thanopoulou AC, Roussi-Penesi DP. Maximal post-prandial triglyceride increase reflects post-prandial hypertriglyceridaemia and is associated with the insulin resistance syndrome. Diabet Med. 2001 Jan;18(1):32-9. doi: 10.1046/j.1464-5491.2001.00386.x. PMID 11168339
- [Background] Carstensen M, Thomsen C, Hermansen K. Incremental area under response curve more accurately describes the triglyceride response to an oral fat load in both healthy and type 2 diabetic subjects. Metabolism. 2003 Aug;52(8):1034-7. doi: 10.1016/s0026-0495(03)00155-0. PMID 12898469
- [Background] Mohanlal N, Holman RR. A standardized triglyceride and carbohydrate challenge: the oral triglyceride tolerance test. Diabetes Care. 2004 Jan;27(1):89-94. doi: 10.2337/diacare.27.1.89. PMID 14693972